CLINICAL TRIAL: NCT03393481
Title: A Multicenter, Randomized, Open-label, Blinded Endpoint Evaluation, Active-controlled Phase 2 Study to Compare the Efficacy and Safety of s.c. MAA868 Versus s.c. Enoxaparin in Adult Patients Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Prevention of Thromboembolic Events in Total Knee Replacement Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial cancelled before First Patient First Visit (no patient enrolled)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMAA868A2201; 2017-002925-39 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Thrombotic Disorders
Keywords: biologic,; venous thromboembolism,; unilateral knee arthroplasty
MeSH Terms: conditions — Venous Thromboembolism | interventions — MAA868; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label, blinded endpoint assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAA868 dose 1 (Experimental): MAA868 dose 1, single administration, subcutaneous
  Interventions: Drug: MAA868
- MAA868 dose 2 (Experimental): MAA868 dose 2, single administration, subcutaneous
  Interventions: Drug: MAA868
- Enoxaparin (Active Comparator): Enoxaparin 40mg, once daily (o.d.) for 10 days
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: MAA868 — MAA868 dose 1 and dose 2, single administration, subcutaneous,
  Arms: MAA868 dose 1; MAA868 dose 2
Drug: Enoxaparin — Enoxaparin 40 mg, o.d X 10 days
  Arms: Enoxaparin

SUMMARY:
The purpose of the study is to find out whether MAA868, is able to prevent blood clots following your medical condition (surgery for knee replacement)

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective unilateral total knee arthroplayts (TKA)
* Willing to comply with study requirements including bilateral venography at Day 12 ± 2 days
* Body weight between 50 kg and 130 kg inclusive.
* Normal aPTT, PT, INR at screening

Exclusion Criteria:

History of arterial or venous thromboembolism; abnormally extended primary or secondary bleeding after trauma or intervention, stroke, transient ischemic attack or traumatic or non-traumatic intracranial bleed; bleeding disorder; MI or unstable angina pectoris within 12 months of the screening; Uncontrolled hypertension (SBP/DBP ≥ 150/95 mmHg at the screening).

Medications that increase the risk of bleeding, including antiplatelet (such as aspirin), anticoagulant and fibrinolytic agents; eGFR < 60 mL/min/1.73m2; Poorly controlled diabetes (HbA1C >10%); Liver dysfunction (ALT/AST >3 xULN or TBL >2 x ULN); BMI ≥ 40 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-03 (Estimated); Primary Completion 2020-01-08 (Estimated); Study Completion 2020-04-17 (Estimated)

PRIMARY OUTCOMES:
Number of patients with confirmed composite endpoint | Day 14
  Occurrence of confirmed composite endpoint of asymptomatic deep vein thrombosis (DVT), confirmed symptomatic venous thromboembolic events (VTE), fatal pulmonary embolism (PE) or unexplained death

SECONDARY OUTCOMES:
Number of patients with composite bleeding | Day 1 to Day 50
  Occurrence of confirmed composite endpoint of major bleeding and clinically relevant non-major (CRNM) bleeding events
Number of patients with composite venous thromboembolic events (VTE) | Day 1 to Day 110
  Occurrence of confirmed composite endpoint of asymptomatic deep vein thrombosis (DVT), Confirmed symptomatic venous thromboembolic events (VTE), fatal pulmonary embolism (PE) or unexplained death

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com